CLINICAL TRIAL: NCT03625921
Title: Effects of a Powered Ankle-Foot Prosthesis and Device-Specific Physical Therapy on Function and Pain for Individuals Living With Transfemoral Limb Loss
Brief Title: Transfemoral Powered Foot and Physical Therapy Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Maikos, Director, VISN 2 Gait and Motion Analysis Laboratory, VA New York Harbor Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB #01643; CDMRP-OP160073 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2018-06-05; First posted 2018-08-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Lower Extremity Problem; Prosthesis User
Keywords: Physical Therapy; Powered Prosthesis; Biomechanical outcomes
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Powered device with physical therapy (Experimental): Subjects will be fitted with a powered ankle-foot prosthesis (Ottobock emPOWER) and provided an intensive device-specific physical therapy (PT) intervention. The subjects will complete, on average, 8 PT training sessions lasting 30 - 45 minutes each. The subjects will also be provided with a home exercise program.
  Interventions: Behavioral: Powered device with physical therapy
- Powered device with standard of practice (Active Comparator): Subjects will be fitted with a powered ankle-foot prosthesis (Ottobock emPOWER) and provided the current standard of practice training for use of this powered prosthesis. The prosthetist will confirm a stable and comfortable alignment and educate the subject on proper home usage. Next, the subject will undergo a 45 - 60 minute training with a physical therapist that is characteristic of the current standard of practice.
  Interventions: Behavioral: Powered device with standard of practice

INTERVENTIONS:
Behavioral: Powered device with physical therapy — Subjects will be fit with a powered prosthesis (Ottobock emPOWER) and enrolled in a device-specific physical therapy (PT) program.
  Arms: Powered device with physical therapy
Behavioral: Powered device with standard of practice — Subjects will be fit with a powered prosthesis (Ottobock emPOWER) and enrolled in the current standard of practice training, which includes basic device education and prosthetic training.
  Arms: Powered device with standard of practice

SUMMARY:
Individuals living with Transfemoral Amputation, enrolled equally at the Veterans Affairs New York Harbor Healthcare System (VANYHHS) and Walter Reed National Military Medical Center (WRNMMC), will be fit with a powered ankle-foot prosthesis. All subjects will undergo a full gait analysis, functional measures, neurocognitive/cognitive, and pain assessment at baseline utilizing their current passive prosthesis. Subjects will then be randomly assigned into 2 equal groups: Powered device with an 8-session intensive, device-specific PT intervention (Group A); or powered device with current standard of practice (Group B), with includes basic device education, but no PT intervention. Subjects in Group A will undergo a 4-week PT-based intervention, which will isolate the contribution of device specific effects from rehabilitation effects. Group B will receive the current standard of practice, which does not include any formal rehabilitation. All users will undergo a full gait analysis, functional measures, neurocognitive/cognitive, and pain assessment after 4- and 8-weeks of use.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral TFA, any etiology
* Experienced (> 6 months) microprocessor knee user
* Less than or equal to 8 amputation related physical therapy sessions in the previous 6 months
* At least 18 y.o.
* High K2 or above ambulator
* Able to walk a minimum of 30 m without an assistive device
* Able to walk on treadmill for 5 minutes at self-selected speed with or without use of handrails

Exclusion Criteria:

* Inability to tolerate wearing of a socket or a poorly fitting socket
* Condition of intact limb prohibits prosthesis use (ulcers, sores, skin breakdown, burns, poor skin coverage, contractures, and severe heterotopic ossification)
* The length of the residual limb prohibits socket/device fitting
* Cognitive deficits or a mental health pathology limiting the ability to participate fully in the study or any deficit deemed by the PI to be detrimental to the completion of the study
* Significant comorbidity, which would interfere with the study (for example: neuropathy, uncontrolled diabetes, receiving dialysis, have insensate feet or severe phantom pain or a history of skin ulcers)
* Severe circulatory problems including peripheral vascular disease and pitting edema
* Pregnant women in the 2nd trimester or beyond or women who will be in the 2nd trimester within the enrollment period. This will be determined by asking the participant if she is pregnant or if they believe they may be pregnant. The question will only be asked at inclusion, as biomechanical changes will only be impacted if the woman is in the 2nd or 3rd trimester, and will not be impacted if the participant becomes pregnant while in the study.
* Weigh more than 287 pounds at screening
* Use of non-prescribed opioids or over-use of any prescription drugs
* Major upper limb amputation
* Currently uses a powered ankle-foot prosthesis as a primary prosthesis or used a powered ankle-foot device as a primary prosthesis in the previous 6 months
* Any cardio-pulmonary, metabolic or integumentary diagnosis where walking for 15 minutes is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Evaluation between PT and non-PT groups | Baseline, Week 4, and Week 8
  Biomechanical evaluation of gait with 3D motion capture while the individual is walking at several different speeds.
Change in 6 minute walk test between PT and non-PT groups | Baseline, Week 4, and Week 8
  The 6-minute walk test measures the distance an individual can walk in 6 minutes without help or encouragement.
Change in AmpPro between PT and non-PT groups | Baseline, Week 4, and Week 8
  The AmpPro is a 21-item instrument designed to measure basic prosthetic mobility of individuals with lower extremity amputation.
Change in the CHAMP between PT and non-PT groups | Baseline, Week 4, and Week 8
  The Comprehensive High-Level Activity Mobility Predictor (CHAMP) is a 4-item, more advanced instrument to measure prosthetic mobility for individuals in this study that scored > 38 on the AmpPro
Change from Baseline in Serial Subtraction at Week 4 and Week 8 | Baseline, Week 4, and Week 8
  Serial Subtraction is a cognitive test where participants are given a random 3 digit number and are asked to subtract by 3s while they walk for 1 minute on a treadmill at a comfortable walking speed. Total number of errors will be documented. Serial subtraction will be performed at baseline using their current prosthetic foot and again at 4- and 8-weeks utilizing the powered prosthesis.
Change from Baseline in COWAT at Week 4 and Week 8 | Baseline, Week 4, and Week 8
  The Controlled Oral Word Association Test (COWAT) is a cognitive test where participants are asked to list as many words as they can think of beginning with a certain letter while walking for 1 minute on a treadmill at a comfortable speed. The participants will complete 3 rounds (3 letters). The total number of unique words for each letter will be documented. COWAT will be performed at baseline using their current prosthetic foot and again at 4- and 8- weeks utilizing the powered prosthesis.
Change from Baseline in Category Test at Week 4 and Week 8 | Baseline, Week 4, and Week 8
  The Category Test is a cognitive test where participants are asked to list as many words as they can think of belonging to a certain category while walking for 1 minute on a treadmill at a comfortable speed. The total number of unique words for the category will be documented. The category test will be performed at baseline using their current prosthetic foot and again at 4- and 8- weeks utilizing the powered prosthesis.
Change from Baseline in CNS Vital Signs at Week 8 | Baseline and Week 8
  The CNS Vital Signs is a computerized neurocognitive assessment that assess 5 domains: memory, psychomotor speed, reaction time, complex attention, and cognitive flexibility. Participants will complete the online platform independently.

SECONDARY OUTCOMES:
Change in Prosthetic Evaluation Questionnaire (PEQ) scores between PT and non-PT groups | Baseline, Week 4, and Week 8
  The PEQ is a self-report Visual Analog Scale questionnaire for persons with lower limb amputations who use a prosthesis. It consists of 9 validated subscales. They are used to evaluate the prosthesis and life with the prosthesis. Most questions in the PEQ use a visual analog scale format. Each visual analog scale is scored as a continuous numerical variable measured as the distance in millimeters from the left endpoint of the line to the point at which the respondent's mark crosses the line. Each line is 100 mm long and is always measured from the left (0-100). The questions are all worded so that a higher number (toward the right) will correspond with a more positive response. Subscale scores are calculated by computing the average (arithmetic mean) of all the questions which make up that particular scale. Only subscales are calculated. A total combined score is not calculated.
Change in Promis Pain Interference levels between PT and non-PT groups | Baseline, Week 4, and Week 8
  The Promis Pain Interference Scale is an 8-item self-report measure of pain interference over the last 7 days. There are 5 potential answers ranging from "not at all" to "very much" for participants to check off. Participants are only allowed to check off one answer per question.
Change in Quality of Life scores between PT and non-PT groups | Baseline, Week 4, and Week 8
  The Quality of Life Scale is a single item visual analog scale used to measure the participants' quality of life over the past four weeks or since their last visit. The visual analog scale is scored as a continuous numerical variable measured as the distance in millimeters from the left endpoint of the line to the point at which the respondent's mark crosses the line. The line is 100 mm long and is always measured from the left (0-100). On the left side of the scale (0 mm) it says "worst possible quality of life". On the right side of the scale (100 mm) it says "ideal quality of life, so the higher the score the more positive the response.
Change in Prosthetic Evaluation Questionnaire-Addendum (PEQ-A) 4 Week responses between PT and non-PT groups | Baseline, Week 4, and Week 8
  The PEQ-A 4 Weeks is a free response 2-item questionnaire in which the participant is asked about any falls and/or stumbles over the last four weeks or since his or her last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Maikos, PhD, Principal Investigator — Director, VISN 2 Gait and Motion Analysis Laboratory
Locations (1):
- VA New York Harbor Healthcare System, New York, New York, United States

REFERENCES:
- [Derived] Maikos JT, Pruziner AL, Hendershot BD, Herlihy DV, Chomack JM, Hyre MJ, Phillips SL, Sidiropoulos AN, Dearth CL, Nelson LM. Effects of a Powered Ankle-Foot Prosthesis and Physical Therapy on Function for Individuals With Transfemoral Limb Loss: Rationale, Design, and Protocol for a Multisite Clinical Trial. JMIR Res Protoc. 2024 Jan 26;13:e53412. doi: 10.2196/53412. PMID 38277197